CLINICAL TRIAL: NCT07365384
Title: Comparison of Pelvic-Free and Pelvic-Restricted Robot-Assisted Gait Training on Walking Pattern, Balance, and Fear of Falling After Stroke
Brief Title: Pelvic-Restricted vs. Pelvic-Free Robot-Assisted Gait Training in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meltem Gunes Akinci (Other)
Responsible Party: Sponsor-Investigator, Meltem Gunes Akinci, Assistant Professor of Physical Medicine and Rehabilitation, Pamukkale University, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-60116787-020-690593
Record Dates: First submitted 2025-09-26; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Hemiplegia; Gait Disorder, Sensorimotor; Balance Impairment; Fear of Falling
MeSH Terms: conditions — Stroke; Hemiplegia; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic-Free Robot-Assisted Gait Training + Conventional Rehabilitation (Experimental): Participants will receive 8 sessions of pelvic-free robot-assisted gait training with RoboGait® (2 sessions per week for 4 weeks) in addition to conventional rehabilitation (5 sessions per week for 4 weeks).
  Interventions: Device: RoboGait® Pelvic-Free Mode; Other: Conventional Rehabilitation
- Pelvic-Restricted Robot-Assisted Gait Training + Conventional Rehabilitation (Active Comparator): Participants will receive 8 sessions of pelvic-restricted robot-assisted gait training with RoboGait® (2 sessions per week for 4 weeks) in addition to conventional rehabilitation (5 sessions per week for 4 weeks).
  Interventions: Device: RoboGait® Pelvic-Restricted Mode; Other: Conventional Rehabilitation

INTERVENTIONS:
Device: RoboGait® Pelvic-Free Mode — Robot-assisted gait training using the RoboGait® system in pelvic-free mode. Participants receive 8 sessions (2 per week for 4 weeks) in addition to conventional rehabilitation.
  Arms: Pelvic-Free Robot-Assisted Gait Training + Conventional Rehabilitation
Device: RoboGait® Pelvic-Restricted Mode — Robot-assisted gait training using the RoboGait® system in pelvic-restricted mode. Participants receive 8 sessions (2 per week for 4 weeks) in addition to conventional rehabilitation.
  Arms: Pelvic-Restricted Robot-Assisted Gait Training + Conventional Rehabilitation
Other: Conventional Rehabilitation — Standard physiotherapy program consisting of 20 sessions (5 per week for 4 weeks) focused on mobility, strengthening, and functional training. Applied to all participants in both groups.

SUMMARY:
This randomized controlled clinical trial aims to compare the effects of pelvic-free versus pelvic-restricted robot-assisted gait training (RAGT) on gait pattern, balance, and fear of falling in stroke patients. Stroke survivors often experience gait impairments, reduced balance, and fear of falling, which limit independence and quality of life. Conventional physiotherapy requires high intensity and repetition but is restricted by therapist capacity. Robotic gait systems provide intensive, repetitive, and safe training; however, most limit pelvic motion, potentially disrupting natural gait patterns and balance strategies.

A total of 36 participants with chronic stroke (≥6 months post-stroke, age ≥18 years, hemiplegic gait disorder, Functional Ambulation Category ≥2) will be randomized into two groups: (1) pelvic-free RAGT plus conventional rehabilitation, or (2) pelvic-restricted RAGT plus conventional rehabilitation. Interventions will consist of 8 RAGT sessions (twice weekly) and 20 conventional rehabilitation sessions (five times weekly) over 4 weeks.

Primary outcomes include gait analysis parameters (gait speed, step length, cadence, temporal symmetry index) and clinical measures such as the Berg Balance Scale, Functional Ambulation Category, Motricity Index (lower limb), and Falls Efficacy Scale-International. Assessments will be performed at baseline and after 4 weeks of treatment.

The study hypothesizes that pelvic-free RAGT will improve gait symmetry, balance, and reduce fear of falling more effectively than pelvic-restricted training. Results are expected to provide evidence supporting the integration of pelvic-free robotic gait systems into post-stroke rehabilitation to enhance functional recovery and patient confidence

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of stroke more than 6 months prior
* Presence of hemiplegia-related gait disorder
* Functional Ambulation Category (FAC) score ≥ 2
* Ability to walk independently prior to stroke

Exclusion Criteria:

* Severe cognitive or communication impairment
* Movement limitations due to joint contracture or deformity
* Presence of open wounds or pressure ulcers
* Uncontrolled hypertension or orthostatic hypotension
* Severe cardiovascular disease, heart failure, cancer, or serious pulmonary disease
* High risk of fracture due to severe osteoporosis
* Gait impairment caused by lower extremity musculoskeletal disorders
* Severe psychosis/neurosis
* Modified Ashworth Scale > 3 in the lower extremities (severe spasticity)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | Baseline (T0) and 4 weeks post-intervention (T1)
  14-item scale assessing static and dynamic balance, scored 0-56 (higher scores indicate better balance).
Gait Speed | Baseline (T0) and 4 weeks post-intervention (T1)
  Gait speed will be assessed using the Zebris FDM-T treadmill system and expressed in meters per second (m/s).
Step Length | Baseline (T0) and 4 weeks post-intervention (T1)
  Step length will be measured with the Zebris FDM-T treadmill system and reported in centimeters (cm).
Cadence | Baseline (T0) and 4 weeks post-intervention (T1)
  Cadence will be recorded using the Zebris FDM-T treadmill system and expressed in steps per minute.
Double Support Time | Baseline (T0) and 4 weeks post-intervention (T1)
  Double support time will be assessed with the Zebris FDM-T treadmill system and expressed as percentage (%) of the gait cycle.
Temporal Symmetry Index | Baseline (T0) and 4 weeks post-intervention (T1)
  Temporal symmetry index will be calculated from gait analysis with the Zebris FDM-T treadmill system and expressed as a percentage (%).

SECONDARY OUTCOMES:
Functional Ambulation Category (FAC) | Baseline (T0) and 4 weeks post-intervention (T1)
  6-level scale (0-5) evaluating functional walking ability, from non-functional ambulation to independent walking.
Motricity Index - Lower Limb | Baseline (T0) and 4 weeks post-intervention (T1)
  Assesses motor function of the paretic lower limb (score range 0-99)
Falls Efficacy Scale-International (FES-I) | Baseline (T0) and 4 weeks post-intervention (T1)
  Self-reported questionnaire evaluating fear of falling during daily activities (higher scores indicate greater fear).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee J, Chun MH, Seo YJ, Lee A, Choi J, Son C. Effects of a lower limb rehabilitation robot with various training modes in patients with stroke: A randomized controlled trial. Medicine (Baltimore). 2022 Nov 4;101(44):e31590. doi: 10.1097/MD.0000000000031590. PMID 36343085
- [Result] Aurich-Schuler T, Gut A, Labruyere R. The FreeD module for the Lokomat facilitates a physiological movement pattern in healthy people - a proof of concept study. J Neuroeng Rehabil. 2019 Feb 6;16(1):26. doi: 10.1186/s12984-019-0496-x. PMID 30728040
- [Result] Alingh JF, Weerdesteyn V, Nienhuis B, van Asseldonk EHF, Geurts ACH, Groen BE. Immediate after-effects of robot-assisted gait with pelvic support or pelvic constraint on overground walking in healthy subjects. J Neuroeng Rehabil. 2019 Mar 15;16(1):40. doi: 10.1186/s12984-019-0506-z. PMID 30876445